CLINICAL TRIAL: NCT03783221
Title: Factors That Determine the Responses to Meal Ingestion: Effect of Previous Diet
Brief Title: Effect of Previous Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PR(AG)338/2016J
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2018-12

CONDITIONS: Healthy
Keywords: meal ingestion; diet; postprandial responses; hedonic sensations; homeostatic sensations; intestinal gas production
MeSH Terms: interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fat diet (Experimental)
  Interventions: Other: High-fat diet
- High-residue diet (Active Comparator)
  Interventions: Other: High-residue diet

INTERVENTIONS:
Other: High-fat diet — The high-fat diet (51% fat, 27% carbohydrates, 21% proteins and 4.7 g fiber) will be administered for two weeks..
  Arms: High-fat diet
Other: High-residue diet — The high-residue diet (19% fat, 62% carbohydrates, 16% proteins and 54.2 g fiber) will be administered for two weeks.
  Arms: High-residue diet

SUMMARY:
Meal ingestion induces digestive responses associated to homeostatic and hedonic sensations. The responses to meal ingestion are modulated by conditioning factors. Single-centre, cross-over, random, open label study comparing the effect of a high-fat/low-residue diet versus low-fat/high residue diet on the responses to meal ingestion. In 20 healthy subjects each diet will be administered during 2 weeks in random order; each diet will be preceded by 2 weeks washout, balanced diet. The aim of the study is to compare the effects of each diet on the responses to comfort and flatulogenic meals, intestinal gas production and digestive sensations.

ELIGIBILITY:
Inclusion Criteria:

* non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Change in digestive well-being induced by comfort meal | 1 day
  Change in digestive well-being measured by a 10 cm scale graded from -5 (extremely unpleasant sensation) to +5 (extremely pleasant sensation) in response to comfort meal during high-fat versus high-residue diet by repeated measures ANCOVA.

SECONDARY OUTCOMES:
Change in fullness sensation induced by comfort meal | 1 day
  Change in fullness sensation measured by a 10 cm scale graded from 0 (not at all) to 10 (very much) in response to comfort meal during high-fat versus high-residue diet by repeated measures ANCOVA.
Change in mood induced by comfort meal | 1 day
  Change in mood measured by a 10 cm scale graded from -5 (negative) to +5 (positive) in response to comfort meal during high-fat versus high-residue diet by repeated measures ANCOVA.
Change in hunger/satiety induced by comfort meal | 1 day
  Change in hunger/satiety measured by a 10 cm scale graded from -5 (extremely hungry) to +5 (completely satiated) in response to comfort meal during high-fat versus high-residue diet by repeated measures ANCOVA.
Intestinal gas evacuation in response to a flatulogenic meal. | 1 day
  Volume of intestinal gas evacuation per anus measured during 4 hours after ingestion of a flatulogenic meal during high-fat versus high-residue diet.
Intestinal gas production | 2 days
  Number of daytime anal gas evacuations measured by an event marker. Participants will be instructed to carry the event marker during daytime and to register every passage of gas per anus for the last two days during high-fat versus high-residue diet.
Sensation of flatulence | 2 days
  Sensation of flatulence measured by a 10 cm scale graded from 0 (not at all) to 10 (very much) for the last two days during high-fat versus high-residue diet.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Pribic T, Azpiroz F. Biogastronomy: Factors that determine the biological response to meal ingestion. Neurogastroenterol Motil. 2018 Jul;30(7):e13309. doi: 10.1111/nmo.13309. Epub 2018 Feb 2. PMID 29392797